CLINICAL TRIAL: NCT01798862
Title: The Effect of Endometrial Injury on IVF Outcome Parameters in Patients With Repeated Implantation Failures
Brief Title: Endometrial Injury and IVF Outcome Parameters in Patients With Failed IVF Cycles
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Siristatidis Charalampos, MD, PhD, Assistant Professor in Obstetrics and Gynecology / Assisted Reproduction, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 121212
Record Dates: First submitted 2013-02-19; First posted 2013-02-26 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Repeated Implantation Failures
Keywords: Failed IVF cycles; IVF outcome parameters; endometrial injury; hysteroscopy; pipelle sampling; Repeated implantation failures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endometrial injury by hysteroscopy or pipelle sapling (Experimental): Endometrial Sampling by pipelle or hysteroscopy performed once between 6th to 10th day in the cycle prior to the fresh IVF/ ICSI cycle.
  Interventions: Procedure: Endometrial injury by hysteroscopy or pipelle sampling
- COH for IVF without hysteroscopy or pipelle sampling (Active Comparator): Procedure: COH for IVF Both GnRH agonists (long, starting at day 2 or 21) with triptorelin acetate 0.1 mg (Gonapeptyl daily) and antagonists with ganirelix 0.25mg (Orgalutran) or cetrorelix 0.25mg (Cetrotide) protocols will be used; for ovarian stimulation both recombinant FSH ( Puregon) and human menopausal gonadotrophin ( Menopur) will be used. Ovarian response will be monitored by ultrasonography, oocyte retrieval will be performed 36-38 hours after the Hcg triggering and for luteal phase support 600 mg progesterone tablets ( Utrogestan) will be applied.
  Interventions: Procedure: Proceed to COH directly

INTERVENTIONS:
Procedure: Endometrial injury by hysteroscopy or pipelle sampling
  Arms: Endometrial injury by hysteroscopy or pipelle sapling
Procedure: Proceed to COH directly
  Arms: COH for IVF without hysteroscopy or pipelle sampling

SUMMARY:
The iatrogenic induction of local endometrial injury caused through hysteroscopy or pipelle sampling in the preceding non- transfer cycle improves the IVF outcome parameters in patients with previous IVF failures.

DETAILED DESCRIPTION:
Endometrial injury was preformed either through hysteroscope during office hysteroscopy through the non touch technique or through pipelle biopsy in the early follicular phase (days 5 to 9) in the preceding cycle of the IVF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Personal history of 2 or more failed IVF/ICSI cycles (RIF)
* Age</= 42 years
* Good response with good quality embryos in previous attempts (>2)

Exclusion Criteria:

* Personal history of endometrial tuberculosis/ antituberculous treatment
* Sonographically detected hydrosalpinges
* Intramural fibroids distorting the endometrial cavity, submucous myomas or Asherman's syndrome
* Thrombophilia

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
positive bHCG rate | through study completion, an average of 2 years

SECONDARY OUTCOMES:
clinical pregnancy rate | 2 years
live birth rate | 2 years
Ectopic pregnancy rate | 2 years
Miscarriage rate | 2 years
Ongoing pregnancy rate | 2 years
Pregnancy complications (preterm birth, placental abnormalities, bleeding throughout pregnancy, pregnancy related hypertensive disorders, IUGR and SGA) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kreatsa, MD/PhD, Principal Investigator — National and Kapodistrian University of Athens; Charalampos Siristatidis, MD, PhD, Principal Investigator — National Kapodistrian University of Athens
Locations (2):
- Greece (2):
  - Assisted Reproduction Unit 3rd Department of Obstetrics & Gynecology, Attikon University Hospital, Athens, Attica
  - Assisted Reproduction Unit, Alexandroupoli, Thrace

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Baum M, Yerushalmi GM, Maman E, Kedem A, Machtinger R, Hourvitz A, Dor J. Does local injury to the endometrium before IVF cycle really affect treatment outcome? Results of a randomized placebo controlled trial. Gynecol Endocrinol. 2012 Dec;28(12):933-6. doi: 10.3109/09513590.2011.650750. Epub 2012 Sep 3. PMID 22943664
- [Result] Karimzadeh MA, Ayazi Rozbahani M, Tabibnejad N. Endometrial local injury improves the pregnancy rate among recurrent implantation failure patients undergoing in vitro fertilisation/intra cytoplasmic sperm injection: a randomised clinical trial. Aust N Z J Obstet Gynaecol. 2009 Dec;49(6):677-80. doi: 10.1111/j.1479-828X.2009.01076.x. PMID 20070722
- [Result] Narvekar SA, Gupta N, Shetty N, Kottur A, Srinivas M, Rao KA. Does local endometrial injury in the nontransfer cycle improve the IVF-ET outcome in the subsequent cycle in patients with previous unsuccessful IVF? A randomized controlled pilot study. J Hum Reprod Sci. 2010 Jan;3(1):15-9. doi: 10.4103/0974-1208.63116. PMID 20607003
- [Result] El-Toukhy T, Sunkara S, Khalaf Y. Local endometrial injury and IVF outcome: a systematic review and meta-analysis. Reprod Biomed Online. 2012 Oct;25(4):345-54. doi: 10.1016/j.rbmo.2012.06.012. Epub 2012 Jun 26. PMID 22885017
- [Result] Potdar N, Gelbaya T, Nardo LG. Endometrial injury to overcome recurrent embryo implantation failure: a systematic review and meta-analysis. Reprod Biomed Online. 2012 Dec;25(6):561-71. doi: 10.1016/j.rbmo.2012.08.005. Epub 2012 Sep 12. PMID 23063812